CLINICAL TRIAL: NCT01970943
Title: Molecular and Functional PET-fMRI Measures of Analgesia in Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, David Borsook, David Borosook, MD, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AT007530-01; R21AT007530-01 (NIH)
Record Dates: First submitted 2013-05-23; First posted 2013-10-28 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Migraine; Healthy
Keywords: migraine, headache, episodic, chronic, pain
MeSH Terms: conditions — Migraine Disorders; Headache; Recurrence; Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): PET-fMRI investigation on healthy subjects and patients with migraine. No drug condition.
- Saline Injection (Placebo) (Placebo Comparator): PET-fMRI investigation on healthy subjects and patients with migraine. Placebo condition.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo will be compared to No Intervention.
  Arms: Saline Injection (Placebo)

SUMMARY:
The placebo effect is a phenomenon that has experienced major advances of its understanding in the last decade. However, mechanisms of placebo analgesia in chronic pain patients have yet to be compared to healthy subjects. The investigators study aims to investigate the magnitude of placebo response and related opioid release in patients that suffer from episodic migraines as compared to healthy controls. In particular, the investigators are looking to map brain activity during placebo analgesia using modern brain imaging techniques such as functional Magnetic Resonance Imaging (fMRI) and Positron Emission Tomography (PET). The investigators hypothesis is that placebo response and the availability of opioid receptors is reduced in chronic migraine patients.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients with aura with acute episodic migraine meeting the IHS Classification ICHD-II criteria, 3-14 migraines per month.
* History of episodic migraine for at least 3 years
* Ages 21-50
* Male or Female
* Right Handed

Matched healthy subjects will also be recruited.

Exclusion Criteria:

* Other significant disease (systemic or CNS)
* Pregnancy
* Claustrophobia
* Weight >235 lbs (limit of MRI table)
* Significant drug including alcohol history (> 7 glasses of alcohol per week)
* Beck Depression Inventory II (BDI-II) score > 25 (moderate to severe depression)
* Any metal implants incompatible with MRI (including dental bridges, crowns, retainers, orthodontic devices e.g. braces, IUDs, aneurysm clips or other devices, tattoos containing metallic ink, cardiac pacemakers, prosthetic hear valves, other prostheses, neurostimulator devices, implanted infusion pumps, exposure to shrapnel or metal filings, cochlear implants, etc.)
* Previous significant research related exposure to ionizing radiation.
* History of allergy or adverse reaction to opioids
* Significant medical history of such as seizure disorder, diabetes, alcoholism, cardiac disease including coronary artery disease, psychiatric problems; drug addiction, respiratory problems, liver disease, etc.
* Positive drug of abuse screen (excluding medications currently prescribed for their clinical condition, e.g. opioids, benzodiazepines, etc.)
* Patients with migraine <72 hours prior to the experiments will not be included to ensure inter-ictal state.
* Opioids or preventative medication such as topiramate, SSRIs etc.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Borsook, MD, Ph.D, Principal Investigator — Boston Children's Hospital
Locations (1):
- Athinoula A. Martinos. Center for Biomedical Imaging, Charlestown, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study design was indeed crossover, but the cross-over was done immediately on the same day. In other words, participants were either scheduled to receive no intervention, and then placed placebo approximately 2 hours later to allow for washout. Or placed placebo first, and then no intervention approximately 2 hours later. No actual drug used.
Groups:
- No Intervention First, Then Placebo: PET-fMRI investigation on healthy subjects and patients with migraine. No drug conditioning and then placebo saline injection.
- Placebo First, Then No Intervention: PET-fMRI investigation on healthy subjects and patients with migraine. Placebo saline injected followed by no drug conditioning.
Period: Overall Study
Arm/Group | No Intervention First, Then Placebo | Placebo First, Then No Intervention
Started | 11 | 12
Completed | 8 | 11
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: healthy subjects and patients with migraine
Groups:
- No Intervention: PET-fMRI investigation on healthy subjects and patients with migraine. No drug condition and placebo (saline IV injection)
Arm/Group | No Intervention
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) 0-10 Pain Rating
Description: This study will investigate how placebo may reduce experimental pain induced by contact heat.
  Patients rate heat stimulus intensity on a 0-10 scale, where 0 is no pain, and 10 is most intense pain possible. Data is reported to the placebo condition.
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'most intense pain possible'. The patient is asked to mark his pain level on the line between the two endpoints.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- No Intervention: PET-fMRI investigation on healthy subjects and patients with migraine. No drug condition and placebo saline injection.
- Placebo: PET-fMRI investigation on healthy subjects and patients with migraine. Placebo saline injection followed by no drug condition.
Arm/Group | No Intervention | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale | 4.3 (2.4) | 7.2 (2.8)

2. Secondary Outcome: Pain Anticipation fMRI BOLD Signal
Description: We imaged the subjects under an MRI scan. All data was collected on a Siemens 3 Tesla MR scanner using a PETcompatible eight-channel head coil. Structural T1 weighted MPRAGE Functional scans were preprocessed using slice timing correction, realignment, normalization, and smoothing (8 mm FWHM Gaussian filter), using SPM12. In each condition (placebo & no drug) subjects underwent four sets of pain anticipation at high and low temperatures (somatosensory control condition). The stimuli were modeled as boxcar time series, with additional regressors for temperature ramp-up, ramp-down, pain rating sequence, and six motion regressors.data were collected for each of the two PET-MR scans. Contrasts analyzed included pain anticipation.
  The values for the 8 sets of anticipation, for both the migraine and the healthy group are combined
Time Frame: 1 day
Population: 9 migraine subjects
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | No Intervention | Placebo
Number analyzed (Participants) | 23 | 23
arbitrary units | 0.5665 (0.8318) | 1.1743 (0.8447)
Statistical Analysis 1: Comparison: No Intervention vs Placebo; Test type: Other; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.6078

3. Secondary Outcome: Pain Stimulation fMRI BOLD Signal
Description: We imaged the subjects under an MRI scan. All data was collected on a Siemens 3 Tesla MR scanner using a PETcompatible eight-channel head coil. Structural T1 weighted MPRAGE Functional scans were preprocessed using slice timing correction, realignment, normalization, and smoothing (8 mm FWHM Gaussian filter), using SPM12. In each condition (placebo & no drug) subjects underwent four sets of pain stimulation at high and low temperatures (somatosensory control condition). The stimuli were modeled as boxcar time series, with additional regressors for temperature ramp-up, ramp-down, pain rating sequence, and six motion regressors.data were collected for each of the two PET-MR scans. Contrasts analyzed included pain stimulation.
  The values for the 8 sets of stimulation, for both the migraine and the healthy group are combined
Time Frame: 1 day
Population: 9 migraine subjects
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | No Intervention | Placebo
Number analyzed (Participants) | 23 | 23
arbitrary units | .5745 (.8224) | 1.1537 (.8326)

4. Secondary Outcome: PET Diprenorphine
Description: We sought to find if endogenous opioid levels and endogenous opioid release induced by placebo administration differentiates between the no intervention first, then placebo group compared to the placebo first, then no intervention group in migraine patients.
Time Frame: 1 day
Population: 9 migraine subjects
Measure: Mean (Standard Deviation); unit: standard uptake value
Arm/Group | No Intervention | Placebo
Number analyzed (Participants) | 23 | 23
standard uptake value | 1.251 (0.259) | 1.214 (0.175)
Statistical Analysis 1: Comparison: No Intervention vs Placebo; Test type: Other; p = .05, t-test, 2 sided; Mean Difference (Final Values) = 0.037786

ADVERSE EVENTS:
Groups:
- Placebo: PET-fMRI investigation on healthy subjects and patients with migraine. Placebo saline injection.
Arm/Group | No Intervention | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No